CLINICAL TRIAL: NCT04760938
Title: Reweaving the Web: Treating Adolescents With CBT and OBH
Brief Title: Treating Adolescents With CBT and OBH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure of comparison group to provide adequate comparison and appropriate comparison
Sponsor: University of New Hampshire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNH-07-8354-01
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Anxiety Disorders; Depressive Disorder; Substance Use Disorders
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Substance-Related Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This is a multi-center, stratified (<$47,000 family income, $47,001-$140,000 family income, >$140,001 family income, with balanced randomization [1:1]), partially-blind, parallel-group study conducted in the United States (7 OBH sites and up to 42 CBT therapists).
Who Masked: Care Provider
Masking Description: Within OBH programs, the field guides are unaware of which participants are study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outdoor Behavioral Healthcare (OBH) (Experimental): Adolescent participants will be asked to complete an intervention in either an OBH program (90 days) or a CBT (12 weeks) program. Parent/guardians and adolescent participants will be asked to complete several surveys before and during the program, and up to one year after.
  Interventions: Behavioral: Outdoor Behavioral Healthcare (OBH)
- Cognitive Behavioral Therapy (CBT) (Experimental): Adolescent participants will be asked to complete an intervention in either an OBH program (90 days) or a CBT (12 weeks) program. Parent/guardians and adolescent participants will be asked to complete several surveys before and during the program, and up to one year after.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Outdoor Behavioral Healthcare (OBH) — Participants in this intervention will participate in one of 7 programs that have been accredited by the Outdoor Behavioral Healthcare Council that specializes in 13-17 year old adolescents experiencing behavioral healthcare issues. Each program works in a unique wilderness setting in various United States National Forests and Parks (e.g., Washington, Oregon, New Mexico, Wisconsin, Utah). The average length of stay in an OBH wilderness program is 90 days, which is a total standard care time of 1,056 hours. All of the OBH programs have been accredited by the Association for Experiential Education Accreditation for Outdoor Behavioral Healthcare programs.
  Other Names: Wilderness Therapy
  Arms: Outdoor Behavioral Healthcare (OBH)
Behavioral: Cognitive Behavioral Therapy (CBT) — The 12-week treatment period will consist of 15 90-minute sessions that will be administered individually. Homework (including reading assignments) are given to encourage your child to practice the techniques learned during the weekly sessions. The total standard of care time for CBT is 22.5 hours of direct treatment hours not including time spent on homework over these twelve weeks. Those therapists that are selected to deliver treatment for the CBT group will be certified by a nationally recognized CBT organization and licensed to work as a therapist in the state where they are providing treatment. Therapy will be delivered in an outpatient setting or through Telehealth.
  Arms: Cognitive Behavioral Therapy (CBT)

SUMMARY:
The purpose of this study is to examine various behavioral, social, and emotional changes that result from engaging in an OBH and CBT treatment program designed for adolescents.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all study participants, including minors and parent/guardians, giving written informed consent will complete a screening survey. The screening survey will support research staff in determining whether participants meet the inclusionary and exclusionary data, including meeting scores on the Youth Outcome Questionnaire and the Revised Children's Anxiety and Depression Scale. If participants are eligible based on preliminary criteria, they undergo a screening interview. If participants are eligible following the screening interview and complete a second informed consent, minors and parents/guardians, they will be randomized in a partially-blind, parallel-group study conducted in the United States (7 Outdoor Behavioral Healthcare programs and up to 42 CBT-licensed therapists).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 13 and 17 years of age
* 5th grade reading level
* For minors, informed assent
* Parental informed consent and adult consent to participate in the study
* Current diagnosis of Depression and/or Anxiety per parent report, parental interview, and score of 65 on the RCADS. Youth with comorbid diagnoses of these listed diagnoses are eligible
* Current secondary diagnosis of Substance Use Disorder (optional)
* Score greater than a 47 on the YoQ-2.0
* Willingness to participate in all aspects of the treatment programs
* Has the ability to carry a pack that is 1⁄4 their body weight

Exclusion Criteria:

* Primary Diagnosis of Substance Use Disorder
* Antisocial Personality
* Level 2 or higher Autism Spectrum
* Schizophrenia
* Actively suicidal
* Eating disorders
* BMI greater than 34
* Diabetic
* Physical ailments or disabilities limiting person from hiking, camping, backpacking
* Specific medications including Anxiolytics/Benzodiazepines, Opiates, or multiple Antipsychotics and Mood Stabilizers
* Youth who have a positive pregnancy test
* Participation in another treatment or intervention study within one year of beginning the study
* Individuals currently suffering from detoxification as a result of drug use in the last five days. If drug use occurs during this time period, the participant must wait until they have achieved five days of substance free behavior. This is done to prevent contraindications of treatment (e.g., interaction between drugs and the environment)
* Currently practicing violent behaviors to self or others within the past year per Parent Report
* Currently experiencing hallucinations (hearing voices or seeing things that are not there)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in statistical and clinical measures on the Youth Outcomes Questionnaire Self-Report (YoQ-SR) at Week 12 | Baseline and Week 12
  The Y-OQ 2.0 has both a parent report global measure of adolescent functioning and an adolescent self-report measure (Y-OQ SR). Both surveys are designed to measure treatment progress for children and adolescents receiving psychological treatment from a parent or caregiver's perspective. Clinical significance is measured by (1) a gain in seven or more points during the clinical trials or (2) a score under 47. The instrument measures overall youth participant functioning that includes six subscales: (a) Intrapersonal Distress, (b) Somatic Symptoms, (c) Interpersonal Relationships, (d) Social Problems, (e) Behavioral Dysfunction, and (f) Critical Items. It is a 64-item parent/guardian report survey designed to assess youth aged 4 to 17 years (Burlingame et al., 2001). Scores for the YoQ-SR range from -16 to +240. The clinical cut-off score is 46. 47 or above represents clinically acute needs.
Change from Baseline in statistical and clinical measures on the Revised Child Anxiety and Depression Scale (RCADS) at Week 12 | Baseline and Week 12
  The Revised Child Anxiety and Depression Scale (RCADS) is a 47-item, youth self-report survey with subscales including: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood (major depressive disorder). It also yields a Total Anxiety Scale (sum of the 5 anxiety subscales) and a Total Internalizing Scale (sum of all 6 subscales). Additionally, The Revised Child Anxiety and Depression Scale - Parent Version (RCADS-P) similarly assesses parent report of youth's symptoms of anxiety and depression across the same six subscales. Scores for the RCADS range from 0 to 141 (47 items on a Likert scale from 0-3). Higher scores signify a worse outcome.
Change from Baseline in statistical and clinical measures on the Family Assessment Device (FAD) at Week 12 | Baseline and Week 12
  The Family Assessment Device (FAD) is a self-report measure that adolescents complete the 10 times (baseline, admission, 5 times during treatment, discharge, 6-months and 12-months post-discharge) and parents complete 5 times (baseline, admission, discharge, 6-months and 12-months post-discharge). The measure consists of seven scales including a General Functioning scale which incorporates items from each of the other scales. The remaining six scales assess the six dimensions of the McMaster Model of Family Functioning which include: (1) Problem Solving, (2) Communication, (3) Roles, (4) Affective Responsiveness, (5) Affective Involvement, and (6) Behavior Control. The FAD has 12 questions scored on a Likert scale from 1-4, resulting in a range of scores from 12 to 48. Higher scores indicate a worse outcome. The clinical cut-off score is 2.0. Scores below 2.0 are normal and scores above 2.0 are clinical.
Change from Baseline in statistical and clinical measures on the Adolescent Alcohol Relapse Coping Questionnaire (ARCQ) at Week 12 | Baseline and Week 12
  The ARCQ is a measure designed to assess temptation coping responses among adolescents with a history of alcohol and drug abuse. The instrument has three factors that represent coping strategies that adolescents utilize when placed in situations that require resisting substance use: (1) cognitive and behavioral problem-solving strategies, (2) self-critical thinking items, & (3) abstinence focused cognitive and behavioral coping items that focus on situational demands of a temptation and the negative consequences of alcohol and drug use.
  The Adolescent Relapse Coping Questionnaire (ARCQ) has a range of scores from 34 to 250. Higher scores indicate stronger endorsement of the particular construct measured.

SECONDARY OUTCOMES:
Change from Baseline in statistical and clinical measures on the Youth Outcomes Questionnaire Self-Report (YoQ-SR) at Week 36 | Baseline and Week 36
  The Y-OQ 2.0 has both a parent report global measure of adolescent functioning and an adolescent self-report measure (Y-OQ SR). Both surveys are designed to measure treatment progress for children and adolescents receiving psychological treatment from a parent or caregiver's perspective. Clinical significance is measured by (1) a gain in seven or more points during the clinical trials or (2) a score under 47. The instrument measures overall youth participant functioning that includes six subscales: (a) Intrapersonal Distress, (b) Somatic Symptoms, (c) Interpersonal Relationships, (d) Social Problems, (e) Behavioral Dysfunction, and (f) Critical Items. It is a 64-item parent/guardian report survey designed to assess youth aged 4 to 17 years (Burlingame et al., 2001). Scores for the YoQ-SR range from -16 to +240. The clinical cut-off score is 46. 47 or above represents clinically acute needs.
Change from Baseline in statistical and clinical measures on the Youth Outcomes Questionnaire Self-Report (YoQ-SR) at Week 60 | Baseline and Week 60
  The Y-OQ 2.0 has both a parent report global measure of adolescent functioning and an adolescent self-report measure (Y-OQ SR). Both surveys are designed to measure treatment progress for children and adolescents receiving psychological treatment from a parent or caregiver's perspective. Clinical significance is measured by (1) a gain in seven or more points during the clinical trials or (2) a score under 47. The instrument measures overall youth participant functioning that includes six subscales: (a) Intrapersonal Distress, (b) Somatic Symptoms, (c) Interpersonal Relationships, (d) Social Problems, (e) Behavioral Dysfunction, and (f) Critical Items. It is a 64-item parent/guardian report survey designed to assess youth aged 4 to 17 years (Burlingame et al., 2001). Scores for the YoQ-SR range from -16 to +240. The clinical cut-off score is 46. 47 or above represents clinically acute needs.
Change from Baseline in statistical and clinical measures on the Revised Child Anxiety and Depression Scale (RCADS) at Week 36 | Baseline and Week 36
  The Revised Child Anxiety and Depression Scale (RCADS) is a 47-item, youth self-report survey with subscales including: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood (major depressive disorder). It also yields a Total Anxiety Scale (sum of the 5 anxiety subscales) and a Total Internalizing Scale (sum of all 6 subscales). Additionally, The Revised Child Anxiety and Depression Scale - Parent Version (RCADS-P) similarly assesses parent report of youth's symptoms of anxiety and depression across the same six subscales. Scores for the RCADS range from 0 to 141 (47 items on a Likert scale from 0-3). Higher scores signify a worse outcome.
Change from Baseline in statistical and clinical measures on the Revised Child Anxiety and Depression Scale (RCADS) at Week 60 | Baseline and Week 60
  The Revised Child Anxiety and Depression Scale (RCADS) is a 47-item, youth self-report survey with subscales including: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood (major depressive disorder). It also yields a Total Anxiety Scale (sum of the 5 anxiety subscales) and a Total Internalizing Scale (sum of all 6 subscales). Additionally, The Revised Child Anxiety and Depression Scale - Parent Version (RCADS-P) similarly assesses parent report of youth's symptoms of anxiety and depression across the same six subscales. Scores for the RCADS range from 0 to 141 (47 items on a Likert scale from 0-3). Higher scores signify a worse outcome.
Change from Baseline in statistical and clinical measures on the Family Assessment Device (FAD) at Week 36 | Baseline and Week 36
  The Family Assessment Device (FAD) is a self-report measure that adolescents complete the 10 times (baseline, admission, 5 times during treatment, discharge, 6-months and 12-months post-discharge) and parents complete 5 times (baseline, admission, discharge, 6-months and 12-months post-discharge). The measure consists of seven scales including a General Functioning scale which incorporates items from each of the other scales. The remaining six scales assess the six dimensions of the McMaster Model of Family Functioning which include: (1) Problem Solving, (2) Communication, (3) Roles, (4) Affective Responsiveness, (5) Affective Involvement, and (6) Behavior Control. The FAD has 12 questions scored on a Likert scale from 1-4, resulting in a range of scores from 12 to 48. Higher scores indicate a worse outcome. The clinical cut-off score is 2.0. Scores below 2.0 are normal and scores above 2.0 are clinical.
Change from Baseline in statistical and clinical measures on the Family Assessment Device (FAD) at Week 60 | Baseline and Week 60
  The Family Assessment Device (FAD) is a self-report measure that adolescents complete the 10 times (baseline, admission, 5 times during treatment, discharge, 6-months and 12-months post-discharge) and parents complete 5 times (baseline, admission, discharge, 6-months and 12-months post-discharge). The measure consists of seven scales including a General Functioning scale which incorporates items from each of the other scales. The remaining six scales assess the six dimensions of the McMaster Model of Family Functioning which include: (1) Problem Solving, (2) Communication, (3) Roles, (4) Affective Responsiveness, (5) Affective Involvement, and (6) Behavior Control. The FAD has 12 questions scored on a Likert scale from 1-4, resulting in a range of scores from 12 to 48. Higher scores indicate a worse outcome. The clinical cut-off score is 2.0. Scores below 2.0 are normal and scores above 2.0 are clinical.
Change from Baseline in statistical and clinical measures on the Adolescent Alcohol Relapse Coping Questionnaire (ARCQ) at Week 36 | Baseline and Week 36
  The ARCQ is a measure designed to assess temptation coping responses among adolescents with a history of alcohol and drug abuse. The instrument has three factors that represent coping strategies that adolescents utilize when placed in situations that require resisting substance use: (1) cognitive and behavioral problem-solving strategies, (2) self-critical thinking items, & (3) abstinence focused cognitive and behavioral coping items that focus on situational demands of a temptation and the negative consequences of alcohol and drug use.
  The Adolescent Relapse Coping Questionnaire (ARCQ) has a range of scores from 34 to 250. Higher scores indicate stronger endorsement of the particular construct measured.
Change from Baseline in statistical and clinical measures on the Adolescent Alcohol Relapse Coping Questionnaire (ARCQ) at Week 60 | Baseline and Week 60
  The ARCQ is a measure designed to assess temptation coping responses among adolescents with a history of alcohol and drug abuse. The instrument has three factors that represent coping strategies that adolescents utilize when placed in situations that require resisting substance use: (1) cognitive and behavioral problem-solving strategies, (2) self-critical thinking items, & (3) abstinence focused cognitive and behavioral coping items that focus on situational demands of a temptation and the negative consequences of alcohol and drug use.
  The Adolescent Relapse Coping Questionnaire (ARCQ) has a range of scores from 34 to 250. Higher scores indicate stronger endorsement of the particular construct measured.

OTHER OUTCOMES:
Explore how youth understand their treatment goals, treatment progress, change process, and potential for long-term change. | Baseline to Week 60
  A series of open-ended questions will be embedded in the survey. Youth complete the questions eight times (admission, five times during treatment, discharge). The questions are designed to explore two basic concepts: 1) How youth understand their treatment goals, treatment progress, change process, and potential for long-term change; and 2) What youth are learning (outcomes), how they are learning (mechanisms), and how they think they will be able to apply their learning outside of the wilderness therapy program (transfer). Youth are instructed to answer the question by writing as much or as little as they like, drawing a picture, creating a poem or sharing lyrics to a song, or using another form to express themselves.
Explore what youth are learning (outcomes), how they are learning (mechanisms), and how they think they will be able to apply their learning outside of the treatment program (transfer). | Baseline to Week 60
  A series of open-ended questions will be embedded in the survey. Youth complete the questions eight times (admission, five times during treatment, discharge). The questions are designed to explore two basic concepts: 1) How youth understand their treatment goals, treatment progress, change process, and potential for long-term change; and 2) What youth are learning (outcomes), how they are learning (mechanisms), and how they think they will be able to apply their learning outside of the wilderness therapy program (transfer). Youth are instructed to answer the question by writing as much or as little as they like, drawing a picture, creating a poem or sharing lyrics to a song, or using another form to express themselves.

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Hampshire, Durham, New Hampshire, United States

REFERENCES:
- See also: Website for study participants to apply to screening survey and obtain study information — https://mypages.unh.edu/unhbehavioralhealthstudy/research